CLINICAL TRIAL: NCT00005214
Title: Epidemiology of Genetic Factors in Lipid Metabolism
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Eric Boerwinkle, Professor, The University of Texas Health Science Center, Houston
Other Study IDs: 1093; R29HL040613 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Genetic variability will be directly assessed by DNA restriction site variability in the apolipoprotein B gene and by measuring the apolipoprotein E polymorphism. These analyses will be carried out on a sample of 75 nuclear families from Nancy France.
  Both fasting and postprandial lipids, lipoproteins, an apolipoproteins will be obtained on a sample of 100 unrelated Mexican-Americans from Laredo, Texas.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the genetics and epidemiology of fasting and postprandial lipid, lipoprotein, and apolipoprotein levels.

DETAILED DESCRIPTION:
BACKGROUND:

Altered plasma lipid, lipoprotein, and apolipoprotein levels are associated with the occurrence of coronary heart disease, non-insulin dependent diabetes, and gallbladder disease. Although there are many other environmental and biological correlates, clinical, epidemiological, and experimental lines of evidence indicate that lipid metabolism has a central role in the development of coronary heart disease. Evidence pointing to the association between measures of lipid metabolism and other chronic diseases is no less compelling. Non-insulin dependent diabetes mellitus exhibits both the diagnostic abnormal carbohydrate utilization, and altered lipid metabolism. The hypothesis that abnormal lipid metabolism may be causally involved in gallbladder disease is suggested by the presence of cholesterol saturated bile several years prior to the onset of clinically definable gallstones.

Biometrical genetic studies have established that a significant proportion of the fasting plasma lipid, lipoprotein, and apolipoprotein levels is attributable to genetic differences among individuals. Although these studies indicate that polygenetic variability is contributing, they do not yield information about specific candidate genes whose products are involved in the metabolism of the phenotype of interest. Recent advances in molecular biology enable one to measure genetic variability at candidate loci for several risk factors for the common chronic diseases. With this information the contribution of specific candidate genes to polygenetic and phenotypic variability can be estimated. Estimating the effects of specific candidate loci will facilitate the investigation of the interaction between genetic and environmental factors. This study focussed on restriction fragment length polymorphisms in and around the apolipoprotein B gene and on the apolipoprotein E protein polymorphism. The apolipoprotein B and apolipoprotein E genes were selected because of their central role in lipid metabolism and interaction with dietary factors.

DESIGN NARRATIVE:

Using data and blood samples from the 75 nuclear families of Nancy, a determination was made of the effects of apolipoprotein B and E genes on fasting levels of total cholesterol and triglycerides, LDL-cholesterol, HDL-cholesterol, HDL2-cholesterol, HDL3-cholesterol, apo A-I, apo-B, apo C-III, and apo-E. Genetic variability was directly assessed by DNA restriction site variability in the apolipoprotein B gene and by measuring the apolipoprotein E polymorphism. Data collected from these families permitted the partitioning of the effects of the apolipoprotein B and E genes from the overall polygenetic and phenotypic variance of the measured lipids, lipoproteins, and apolipoproteins.

Fasting and postprandial lipids, lipoproteins, and apolipoproteins were obtained from 100 Mexican-American women. A determination was made of the effects of apolipoprotein E and B genes, disease status, age, and their interactions on fasting and postprandial lipid metabolism.

ELIGIBILITY:
No eligibility criteria

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Sample of 75 nuclear families from Nancy France. Sample of 100 unrelated Mexican-Americans from Laredo, Texas.
Dates: Start 1988-04; Study Completion 1993-03

REFERENCES:
- [Background] Surguchov AP, Page GP, Smith L, Patsch W, Boerwinkle E. Polymorphic markers in apolipoprotein C-III gene flanking regions and hypertriglyceridemia. Arterioscler Thromb Vasc Biol. 1996 Aug;16(8):941-7. doi: 10.1161/01.atv.16.8.941. PMID 8696957
- [Background] Boerwinkle E, Xiong WJ, Fourest E, Chan L. Rapid typing of tandemly repeated hypervariable loci by the polymerase chain reaction: application to the apolipoprotein B 3' hypervariable region. Proc Natl Acad Sci U S A. 1989 Jan;86(1):212-6. doi: 10.1073/pnas.86.1.212. PMID 2911570
- [Background] Boerwinkle E, Chan L. A three codon insertion/deletion polymorphism in the signal peptide region of the human apolipoprotein B (APOB) gene directly typed by the polymerase chain reaction. Nucleic Acids Res. 1989 May 25;17(10):4003. doi: 10.1093/nar/17.10.4003. PMID 2567503
- [Background] Gueguen R, Visvikis S, Steinmetz J, Siest G, Boerwinkle E. An analysis of genotype effects and their interactions by using the apolipoprotein E polymorphism and longitudinal data. Am J Hum Genet. 1989 Nov;45(5):793-802. PMID 2816943
- [Background] Visvikis S, Chan L, Siest G, Drouin P, Boerwinkle E. An insertion deletion polymorphism in the signal peptide of the human apolipoprotein B gene. Hum Genet. 1990 Mar;84(4):373-5. doi: 10.1007/BF00196239. PMID 2307462
- [Background] Seed M, Hoppichler F, Reaveley D, McCarthy S, Thompson GR, Boerwinkle E, Utermann G. Relation of serum lipoprotein(a) concentration and apolipoprotein(a) phenotype to coronary heart disease in patients with familial hypercholesterolemia. N Engl J Med. 1990 May 24;322(21):1494-9. doi: 10.1056/NEJM199005243222104. PMID 2139920
- [Background] Boerwinkle E, Lee SS, Butler R, Schumaker VN, Chan L. Rapid typing of apolipoprotein B DNA polymorphisms by DNA amplification. Association between Ag epitopes of human apolipoprotein B-100, a signal peptide insertion/deletion polymorphism, and a 3'flanking DNA variable number of tandem repeats polymorphism of the apolipoprotein B gene. Atherosclerosis. 1990 Apr;81(3):225-32. doi: 10.1016/0021-9150(90)90070-y. PMID 1693506
- [Background] Visvikis S, Steinmetz J, Boerwinkle E, Gueguen R, Galteau MM, Siest G. Frequency and effects of the apolipoprotein A-IV polymorphism. Clin Genet. 1990 Jun;37(6):435-41. doi: 10.1111/j.1399-0004.1990.tb03527.x. PMID 2383930
- [Background] Boerwinkle E, Visvikis S, Chan L. Two polymorphisms for amino acid substitutions in the APOA4 gene. Nucleic Acids Res. 1990 Aug 25;18(16):4966. doi: 10.1093/nar/18.16.4966. No abstract available. PMID 2395672
- [Background] de Temmerman P, Visvikis S, Boerwinkle E, Siest G. Study of the sequence tagged site (STS) in the beginning of human apo A4 gene region. Nucleic Acids Res. 1990 Sep 25;18(18):5576. doi: 10.1093/nar/18.18.5576. PMID 2216752
- [Background] Xu CF, Boerwinkle E, Tikkanen MJ, Huttunen JK, Humphries SE, Talmud PJ. Genetic variation at the apolipoprotein gene loci contribute to response of plasma lipids to dietary change. Genet Epidemiol. 1990;7(4):261-75. doi: 10.1002/gepi.1370070405. PMID 1977654
- [Background] Boerwinkle E, Hanis CL, Chan L. A unique length polymorphism in the signal peptide region of the apolipoprotein B gene in Mexican-Americans. Nucleic Acids Res. 1990 Dec 11;18(23):7193. doi: 10.1093/nar/18.23.7193. PMID 2263508
- [Background] Talmud PJ, Boerwinkle E, Xu CF, Tikkanen MJ, Pietinen P, Huttunen JK, Humphries S. Dietary intake and gene variation influence the response of plasma lipids to dietary intervention. Genet Epidemiol. 1992;9(4):249-60. doi: 10.1002/gepi.1370090404. PMID 1356882
- [Background] Shriver MD, Siest G, Boerwinkle E. Length and sequence variation in the apolipoprotein B intron 20 Alu repeat. Genomics. 1992 Oct;14(2):449-54. doi: 10.1016/s0888-7543(05)80240-x. PMID 1427859
- [Background] Boerwinkle E, Leffert CC, Lin J, Lackner C, Chiesa G, Hobbs HH. Apolipoprotein(a) gene accounts for greater than 90% of the variation in plasma lipoprotein(a) concentrations. J Clin Invest. 1992 Jul;90(1):52-60. doi: 10.1172/JCI115855. PMID 1386087
- [Background] Fornage M, Chan L, Siest G, Boerwinkle E. Allele frequency distribution of the (TG)n(AG)m microsatellite in the apolipoprotein C-II gene. Genomics. 1992 Jan;12(1):63-8. doi: 10.1016/0888-7543(92)90407-j. PMID 1733865
- [Background] Lackner C, Boerwinkle E, Leffert CC, Rahmig T, Hobbs HH. Molecular basis of apolipoprotein (a) isoform size heterogeneity as revealed by pulsed-field gel electrophoresis. J Clin Invest. 1991 Jun;87(6):2153-61. doi: 10.1172/JCI115248. PMID 1645755
- [Background] Boerwinkle E, Brown SA, Rohrbach K, Gotto AM Jr, Patsch W. Role of apolipoprotein E and B gene variation in determining response of lipid, lipoprotein, and apolipoprotein levels to increased dietary cholesterol. Am J Hum Genet. 1991 Dec;49(6):1145-54. PMID 1746549
- [Background] Boerwinkle E, Chen SH, Visvikis S, Hanis CL, Siest G, Chan L. Signal peptide-length variation in human apolipoprotein B gene. Molecular characteristics and association with plasma glucose levels. Diabetes. 1991 Nov;40(11):1539-44. doi: 10.2337/diab.40.11.1539. PMID 1936612
- [Background] Hallman DM, Boerwinkle E, Saha N, Sandholzer C, Menzel HJ, Csazar A, Utermann G. The apolipoprotein E polymorphism: a comparison of allele frequencies and effects in nine populations. Am J Hum Genet. 1991 Aug;49(2):338-49. PMID 1867194
- [Background] Mancini FP, Mooser V, Guerra R, Hobbs HH. Sequence microheterogeneity in apolipoprotein(a) gene repeats and the relationship to plasma Lp(a) levels. Hum Mol Genet. 1995 Sep;4(9):1535-42. doi: 10.1093/hmg/4.9.1535. PMID 8541836
- [Background] Carrejo MH, Sharrett R, Patsch W, Boerwinkle E. No association of apolipoprotein A-IV codon 347 and 360 variation with atherosclerosis and lipid transport in a sample of mixed hyperlipidemics. Genet Epidemiol. 1995;12(4):371-80. doi: 10.1002/gepi.1370120405. PMID 8536954
- [Background] Moliterno DJ, Jokinen EV, Miserez AR, Lange RA, Willard JE, Boerwinkle E, Hillis LD, Hobbs HH. No association between plasma lipoprotein(a) concentrations and the presence or absence of coronary atherosclerosis in African-Americans. Arterioscler Thromb Vasc Biol. 1995 Jul;15(7):850-5. doi: 10.1161/01.atv.15.7.850. PMID 7600116
- [Background] de Andrade M, Thandi I, Brown S, Gotto A Jr, Patsch W, Boerwinkle E. Relationship of the apolipoprotein E polymorphism with carotid artery atherosclerosis. Am J Hum Genet. 1995 Jun;56(6):1379-90. PMID 7762561
- [Background] Hallman DM, Visvikis S, Steinmetz J, Boerwinkle E. The effect of variation in the apolipoprotein B gene on plasmid lipid and apolipoprotein B levels. I. A likelihood-based approach to cladistic analysis. Ann Hum Genet. 1994 Jan;58(1):35-64. doi: 10.1111/j.1469-1809.1994.tb00724.x. PMID 8031014
- [Background] Boerwinkle E, Brown S, Sharrett AR, Heiss G, Patsch W. Apolipoprotein E polymorphism influences postprandial retinyl palmitate but not triglyceride concentrations. Am J Hum Genet. 1994 Feb;54(2):341-60. PMID 8304350
- [Background] Moliterno DJ, Lange RA, Meidell RS, Willard JE, Leffert CC, Gerard RD, Boerwinkle E, Hobbs HH, Hillis LD. Relation of plasma lipoprotein(a) to infarct artery patency in survivors of myocardial infarction. Circulation. 1993 Sep;88(3):935-40. doi: 10.1161/01.cir.88.3.935. PMID 8353920